CLINICAL TRIAL: NCT04121260
Title: A Phase 1, Open-label, Multicenter Study of Subcutaneous Delivery of JNJ-54767414 (Daratumumab) in Chinese Subjects With Multiple Myeloma
Brief Title: A Study of Subcutaneous Delivery of JNJ-54767414 in Chinese Participants With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108638; 54767414MMY1010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Daratumumab (Experimental): Participants will receive daratumumab dose 1 subcutaneously (SC) with recombinant human hyaluronidase [rHuPH20] 30,000 units [U] that is 2,000 U/milliliter (U/mL) SC injection once weekly for the first 8 weeks Cycles 1 and 2 (Days 1, 8, 15, and 22 of each week), every 2 weeks Cycles 3 to 6 (Days 1 and 15) or the following 16 weeks and then every 4 weeks from Cycle 7 [Day 1] in subsequent cycles, until disease progression, unacceptable toxicity, or any other reason for discontinuation. Each cycle is 28 days in duration.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Participants will receive dose 1 daratumumab with 30,000 U (2000 U/mL) with rHuPH20 SC injection.
  Other Names: JNJ-54767414

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetic of Daratumumab subcutaneously in Chinese participants with relapsed or refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma (MM) diagnosed according to the International Myeloma Working Group (IMWG) diagnostic criteria
* Participants must have measurable, secretory disease as defined by any of the following:

  1. Serum monoclonal paraprotein (M-protein) level greater than or equal to(>=)1.0 gram/deciliter (g/dL) or >= 0.5 g/dL for Immunoglobulin (Ig) A, IgD, IgE or IgM MM; or
  2. Urine M-protein level >= 200 milligram (mg)/24 hours; or
  3. Serum Ig free light chain (FLC) >= 10 mg/dL and abnormal serum Ig kappa lambda FLC ratio if participant does not have measurable M-protein in serum and urine
* Relapsed or refractory MM after receiving at least 2 prior lines of therapy: Received both, a PI (>=2 cycles or 2 months of treatment) and an IMiD (>=2 cycles or 2 months of treatment)in any order during the course of treatment (except for participants who discontinued either of these treatments due to a severe allergic reaction within the first 2 cycles/months); A "line of therapy" is defined as 1 or more cycles of a planned treatment program, Radiotherapy, bisphosphonate therapy, or a single short course of steroids (that is, less than or equal to equivalent of cumulative dose of dexamethasone 160 mg within 21 days of 1st dose) would not be considered prior lines of therapy
* Response (partial response or better based on investigator's determination of response) to at least 1 prior treatment regimen
* Progressive disease based on investigator's determination of response on or after their last regimen
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Participant has received daratumumab or other anti-CD38 therapies previously
* Participant has received prior antitumor therapy as follows, prior to the first dose of study drug:

  1. Targeted therapy, epigenetic therapy, or treatment with an investigational drug or an invasive investigational medical device within 21 days or at least 5 half-lives, whichever is less;
  2. Monoclonal antibody treatment for multiple myeloma within 21 days;
  3. Cytotoxic therapy within 21 days;
  4. Proteasome inhibitor therapy within 14 days;
  5. Immunomodulatory agent therapy within 7 days;
  6. Radiotherapy within 21 days. However, if the radiation portal covered less than or equal to (<=) 5 percent (%) of the bone marrow reserve, the participant is eligible irrespective of the end date of radiotherapy
* Participant has had a plasmapheresis within 28 days before Cycle 1 Day 1
* Participant has known meningeal or central nervous system involvement of MM
* Concurrent medical condition or disease (example [e.g.], active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious AEs | Up to 2 years
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Maximum Observed Serum Concentration (Cmax) of Daratumumab | Day 1 (2 hours, 12 hours) Cycle 1 (each cycle is of 28 days)
  Cmax is the maximum observed serum concentration.
Serum Trough Concentration (Ctrough) of Daratumumab | At Day 1 Cycle 3 predose concentration (each cycle is of 28 days)
  Ctrough is the observed concentration of daratumumab prior to the next drug administration.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years
  ORR, defined as the percentage of participants with a partial response (PR) or better according to the International Myeloma Working Group (IMWG) response criteria.
Duration of Response (DOR) | Up to 2 years
  DOR, defined as date of onset of first response until date of disease progression or death (according to the IMWG response criteria).
Time to Response | Up to 2 years
  TTR, defined as the time from Cycle 1 Day 1 until onset of first response (according to the IMWG response criteria).
Serum Concentration of Daratumumab and Recombinant Human Hyaluronidase (rHuPH20) (Plasma) Antibodies | Up to 2 years
  Serum levels of antibodies to Daratumumab and rHuPH20 for evaluation of potential immunogenicity will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- China (5):
  - Peking University Third Hospital, Beijing
  - The Third Xiangya Hospital, Central South University, Changsha
  - Nanfang Hospital, Guangzhou
  - Zhongda Hospital,Southeast University, Nanjing
  - Institute of Hematology & Blood Diseases Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] An G, Ge Z, Jing H, Liu J, Yang G, Feng R, Xu Z, Qi M, Wang J, Song J, Zhou W, Sun B, Zhu D, Chen X, Cui C, Qiu L. Subcutaneous daratumumab in Chinese patients with relapsed or refractory multiple myeloma: an open-label, multicenter, phase 1 study (MMY1010). Blood Sci. 2024 May 31;6(3):e00193. doi: 10.1097/BS9.0000000000000193. eCollection 2024 Jul. PMID 38832105